CLINICAL TRIAL: NCT00789620
Title: Effects of Intravenous Lidocaine on Transperitoneal Laparoscopic Urological Surgery: A Prospective, Randomised, Placebo Controlled, Double-blind, Phase III Study
Brief Title: Effects of Intravenous Lidocaine on Transperitoneal Laparoscopic Urological Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Patrick Y Wüthrich MD, Dep. of anesthesiology and pain service, Bern University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KEK_155_08
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Pain; Fatigue
Keywords: intravenous lidocaine; laparoscopic urological surgery; hospital stay; pain; fatigue; length of stay
MeSH Terms: conditions — Pain; Fatigue | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Lidocaine 1% administrated as a bolus of 1.5 mg/kg, then intraoperative 2mg/kg/h and postoperative 1.3mg/kg/h during 24 h
  Interventions: Drug: lidocaine
- 2 (Placebo Comparator): NaCl 0.9% as a bolus 1.5mg/kg, then intraoperative 2mg/kg/h and postoperative 1.3mg/kg/h during 24h
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lidocaine — 1.5 mg/kg as Bolus intraoperative: 2 mg/kg/h postoperative: 1.3mg/kg/h during 24h
  Arms: 1
Drug: placebo — Bolus 0.15 ml/kg NaCl 0.9% NaCl 0.2 ml/kg/h Perfusor NaCl 0.9% 0.13 ml/kg/h Perfusor
  Arms: 2

SUMMARY:
Effective perioperative analgesia is the key to postoperative rehabilitation. An intriguing body of evidence suggests that short-term administration of intravenous lidocaine may produce pain relief that far exceeds both the duration of infusion and the half-life of the drug. When pain relief is provided, concomitant anal-gesic medication can be reduced, side effects from pain relieving medication minimized with a potential for a more rapid postoperative recovery and less complications. IV application of lidocaine should de-crease the duration of bowel dysfunction. We hypothesise that i.v. application of lidocaine in a standard antiarrythmic dose can significantly improve acute rehabilitation after laparoscopic urological surgery and so shorten the hospital stay (primary outcome). We expect that the intraoperative inflammatory response can significantly be reduced.

DETAILED DESCRIPTION:
Effective perioperative analgesia is the key to postoperative rehabilitation. It has been suggested that a decrease in postoperative pain and opioid use ameliorates the return of normal bowel function after general surgery. Conventional analgesic treatment involves the use of intravenous, oral and transdermal formulations of drugs. Repetitive administration is required for sustained pain relief. Common side effects (postoperative nausea and vomiting, postoperative ileus) of these analgesics may have a detrimental effect on postoperative recovery and led to a prolonged hospital stay. An intriguing body of evidence suggests that short-term administration of intravenous lidocaine may produce pain relief that by far exceeds both the duration of the infusion and the half-life of the drug thus reducing concomitant analgesic medication can be reduced and its side effects enabling a more rapid postoperative recovery with less complications. Lidocaine is a commonly used local anesthetic and an antiarrythmic agent. It has been shown to preserve neuroelectric function in animal experiments. Intraoperative administration of lidocaine in a standard antiarrythmic dose has been shown to decrease the occurrence of cognitive dysfunction in the early postoperative period after coronary artery bypass surgery. Lidocaine can induce a significant re-duction of several components of chronic pain in patients with poststroke or spinal cord injury related pain. Sodium channel blockers (e.g. lidocaine) are approved for intravenous administration in the treat-ment of neuropathic pain states. In addition lidocaine has anti-inflammatory properties and preclinical studies have suggested antihyperalgesic effects on the peripheral and central nervous system. Lidocaine decreases the minimum alveolar concentration (MAC) of inhaled anesthetics and has been used clinically to reduce the requirements for other anesthetic drugs. IV application of lidocaine is said to decrease the duration of bowel dysfunction and postoperative pain intensity.

We hypothesise that i.v. application of lidocaine in a standard antiarrythmic dose can significantly improve acute rehabilitation after laparoscopic urological surgery and so shorten the hospital stay. We expect that the intraoperative inflammatory response can significantly be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ASA 1 to 3
* Laparoscopic transperitoneal urological surgery

Exclusion Criteria:

* Liver insufficiency
* Steroid therapy
* Chronic opioid therapy
* Allergy to lidocaine
* Pre-existing disorder of the gastrointestinal tract
* AV-block II-III, sinusbradycardia, heart insufficiency, long QT-syndrome
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Hospital stay | end of hospitalisation

SECONDARY OUTCOMES:
change in pain score | 2 and 4 h postop and 3*/d on day 1 and 2
changes in fatigue score | 2 and 4 h postop and 3*/d on day 1 and 2
PONV | 2 and 4 h postop and 3*/d on day 1 and 2
time to first episode of flatus and defecation | 2 and 4 h postop and 3*/d on day 1 and 2
changes in metabolic and inflammatory responses (cortisol, glc, CRP and procalcitonin) | preoperatively and on day 1 and 2 in the morning

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wüthrich, MD, Principal Investigator — Dep. of Anesthesiology and pain service, Bern University Hospital
Locations (1):
- Dep. of Urology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Wuethrich PY, Romero J, Burkhard FC, Curatolo M. No benefit from perioperative intravenous lidocaine in laparoscopic renal surgery: a randomised, placebo-controlled study. Eur J Anaesthesiol. 2012 Nov;29(11):537-43. doi: 10.1097/EJA.0b013e328356bad6. PMID 22907609